CLINICAL TRIAL: NCT04478747
Title: Women's Apical Pelvic Organ Prolapse Treatment - a Randomized Controlled Trial Comparing Transvaginal and Laparoscopic Mesh Surgery
Brief Title: Transvaginal Mesh vs. Laparoscopic Colposacropexy- Study
Acronym: TVM vs LCSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Camilla Isaksson, Senior consultant, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01072020
Record Dates: First submitted 2020-06-15; First posted 2020-07-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Prolapse, Vaginal Vault
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transvaginal mesh (Active Comparator): BSC mesh (A.M.I., Feldkirch, Austria) is attached to the sacrospinosus ligaments and to the apical part of the vagina.
  Interventions: Procedure: TVM
- Colposacropexy with the apical fixation only (Active Comparator): EndoGYNious (A.M.I.) CSP mesh is attached laparoscopically to the apical part of the vagina.
  Interventions: Procedure: Colposacropexy
- Colposacropexy with the apical and the levator fixation (Active Comparator): EndoGYNious (A.M.I.) CSP mesh is attached laparoscopically to the apical part of the vagina with fixation reaching to the level of the levator planes.
  Interventions: Procedure: Colposacropexy

INTERVENTIONS:
Procedure: TVM — Transvaginal mesh operation using BSC mesh (A.M.I., Feldkirch, Austria)
  Arms: Transvaginal mesh
Procedure: Colposacropexy — Colposacropexy using EndoGYNious mesh (A.M.I., Feldkirch, Austria)
  Arms: Colposacropexy with the apical and the levator fixation; Colposacropexy with the apical fixation only

SUMMARY:
The main objective of the study is to compare subjective efficacy of trans vaginal mesh and laparoscopic colposakropexy (CSP) in women with an apical prolapse. The CSP group is further divided into two sub-groups; one where the mesh fixation is only at the apical part of the vagina, and another where the fixation is also extended to the levator plane.

The secondary outcomes are safety (peri- and post-surgery complications, pain, erosion), objective efficacy (simplified POP-Q), and re-operation rate. Subjective outcome also includes the assessment of sexual satisfaction. Cost-effectiveness is studied by comparing both direct costs and QALYs.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is defined as an anatomical support defect of the pelvic viscera. Women's POP is the descent of uterus or vaginal apex with or without concomitant descent of the anterior (cystocele) or posterior (rectocele) vaginal wall. It is estimated that the lifetime risk of POP surgery in women is approximately 10-13%, the incidence peak being 20-30 years after the first delivery, which is also the most important risk factor for POP. Other risk factors include previous hysterectomy, obesity and genetic factors.

The typical POP symptoms are a feeling of bulge, accompanied with urinary incontinence, defecation problems, and sexual dissatisfaction. First line treatments are conservative, but if they fail, surgery is indicated.

Native tissue repair of the anterior and / or posterior vaginal wall (colporrhaphy anterior / posterior) is commonly the first-line operation. The possible concomitant apical prolapse needs to be suspended which is typically done by either by performing a hysterectomy with shortening and suspension of the sacrouterine ligaments, or by amputation of the cervix with suspension of the cardinale and sacrouterine ligaments (Manchester operation). An unsuspended apical defect will double the relapse rate (20 vs 11%). In most of the apical recurrences mesh is used to achieve sufficient support. The re-operation rate of any POP in Finland is 10.8% .

In mesh operations the apex can be suspended either transvaginally (TVM) by anchoring the mesh to the sacrospinosus ligaments, or by doing a colposacropexy (CSP) where the mesh is attached to the sacrum, mostly via laparoscopy. The CSP techniques vary e.g. the mesh can be attached only apically or also to the levator plane. If needed, colporrhaphies can be done concomitantly.

The use of TVM has decreased due to the FDA-warnings and litigations concerning mainly the risks of erosion and pain. This has lead to withdrawals of mesh products, despite well-conducted clinical studies indicating that in well-chosen women light-weight small TVM is not associated with major complications. Currently, no TVM with good quality clinical data is available. Traditionally, CSP has been considered safer than TVM in regard of erosions and pain, but the data is scarce. Furthermore, CSP has a longer learning-curve and is a more time-consuming operation than TVM, whereas hospital stay is shorter.

To the investigators knowledge, there is only one published study where TVM and CSP has been compared, and in that study a large "covering" TVM was used which was thereafter withdrawn from the market. In addition,in most studies, operation techniques, especially with CSP are not standardized. Therefore, further head-to-head comparisons are needed. The investigators propose a study comparing efficacy and safety when using the TVM or CSP approach in women with an apical defect. The investigators will also evaluate whether, in CSP, apical fixation alone is sufficient, or whether levator plane fixation provide a better outcome.

Study objective:

The main objective of the study is to compare subjective efficacy (PFDI-20, question nro 3; feeling of bulge) between TVM and CSP in women with an apical prolapse. The CSP group is further divided into two sub-groups; one where the mesh fixation is only at the apical part of the vagina, and another where the fixation is also extended to the levator plane.

The secondary outcomes are safety (peri- and post-surgery complications, pain, erosion), objective efficacy (simplified POP-Q), and re-operation rate. Subjective outcome also includes the assessment of sexual satisfaction. Cost-effectiveness is studied by comparing both direct costs and QALYs.

Inclusion criteria:

Age over 18 years and capability to understand the study protocol either in Finnish or Swedish.

Objectively diagnosed symptomatic apical prolapse (leading apical prolapse (points C/D ≥-2) and a history of previous POP operation including hysterectomy.

No need for any other concomitant operations except colporrhaphies and possible prophylactic salpingo-oophorectomy in CSP groups

Exclusion criteria:

A history of previous serious or prolonged pain after any operation. Regular use of systemic corticosteroid medication. Incapability to understand the study protocol.

Groups, procedures, and randomization:

The participants are randomized into three groups:

1. Transvaginal mesh: BSC mesh (A.M.I., Feldkirch, Austria) is attached to the sacrospinous ligaments and to the apical part of the vagina. Briefly, 0,25% Lidocain solution with adrenaline is injected to the anterior vaginal wall and towards the sacrospinous ligaments bilaterally to reduce bleeding and aid dissection. A vertical incision to the anterior vaginal wall is done from a point below the bladder neck to approximately 1cm from the vaginal apex. A full-thickness blunt dissection is done leaving the vaginal fascia laterally, with tunneling to the sacrospinous ligaments. The two arms of the mesh are attached with an i-Stich instrument (A.M.I.) to the sacrospinous ligaments 1-2 cm laterally from the ischial spines. The anterior edge of the mesh is attached to the vaginal fascia with three Monocryl 3-0 sutures. If needed, the mesh may be shortened in length and is so, the removed piece is measured and recorded. The arms of the mesh are set to the stage that the vaginal wall is reduced to its natural position. Complete vaginal wound closure is done with Vicryl 3-0 sutures. A roll of vaginal gauze for compression is applied and foley catheter inserted until the following morning. A single i.v. dose of 1.5g cefuroxime antibiotic is given at the time of anesthesia induction.
2. Colposacropexy with the apical fixation only: PelviGYNious (A.M.I., Feldkirch, Austria) CSP mesh is attached laparoscopically to the apical part of the vagina. Briefly, a single i.v. dose 1.5 g of cefuroxime is administered at the time of the anesthesia induction. The umbilical entry is done optically by a 11 mm trocar and a pneumoperitoneum up to 12 mmHg is created (then lowered to 8 mmHg, if possible, after all trocars are inserted). A five mm trocar is placed to the left lower abdomen, a 11 mm trocar on the left side superior to the previous and a 7.5 mm Airseal trocar to the right lower abdomen. The promontory is visualized and the avascular space is dissected by an advanced energy instrument (Thunderbeat, Olympus). The right ureter, the major vessels and the right hypogastric nerve trunk are identified and avoided during the dissection. Opening of the right pelvic peritoneum is done with dissection of the pararectal space. The posterior vaginal peritoneum is opened below the level of the insertions of the uterosacral ligaments (USL) and the opening is extended to the peritoneum over the left pararectal area. The rectovaginal and the left pararectal spaces are dissected to create a posterior peritoneal flap. Anteriorly, the peritoneum below the vaginal apex is opened and dissected to create an anterior peritoneal flap. A CSP mesh is fixed to the vaginal apex with five non-absorbable Surgilon 2-0 sutures utilizing an extracorporeal knot-tying technique: three in a row to the apex and two to the sides two centimeters posterior to the apex (or alternatively three sutures to the cervix if it is present). A vaginal speculum examination is performed and any sutures penetrating the vaginal mucosa are removed and replaced with new ones. The tension of the mesh is controlled visually via a speculum examination. Anterior and/or posterior colporraphy is introduced at this point if a vaginal wall prolapse exceeding -2 position is seen after tensioning the mesh. The mesh is attached to the promontory with five fasteners (CapSure, Bard). The peritoneum is closed by a running V-Loc™.
3. Colposacropexy with the apical and the levator fixation: PelviGYNious (A.M.I., Feldkirch, Austria) CSP mesh is attached laparoscopically to the apical part of the vagina with fixation reaching to the level of the levator planes. Briefly, the technique is similar to the apical fixation with the following exceptions: the pararectal spaces are dissected deep to the level of the levator ani muscles and the CSP mesh is fixed with 11 sutures (figure) (two to the levator ani muscles, two to the insertions of the USLs and two to the midline of the posterior vaginal wall; the apical fixation is done similar to the former group).

In all groups concomitant colporrhaphies can be conducted. Anterior or posterior colporraphy is done in the following fashion: a 0,25% lidocaine solution containing adrenaline is injected under the anterior or posterior vaginal wall to provide haemostasis and hydrodissection. The vaginal wall is incised and the fascia is separated from the vaginal epithelium using a combination of sharp and blunt dissection. The fascia is plicated using a running 3-0 PDS suture in two layers. Excess vaginal epithelium is excised and the vaginal epithelium is closed with a running 3-0 Vicryl suture.

All the operators have conducted at least ten surgeries with the mesh before taking part into the study.

Power calculation:

The primary outcome is subjective success; defined as the absence of vaginal bulge, i.e. negative response to PDFI-20, question 3 at one-year following the surgery. Previous literature show various results. Altman et al (NEJM 2011) described that this outcome was achieved in 61% of women following a transvaginal mesh surgery. A prospective study by Duraes et al (2019) and Wei et al described an even higher success of 92% to 94%. Laparoscopic CSP has shown a subjective success rate of 91% to 94%. Based on these findings we assumed that the subjective success would be 80% following laparoscopic CSP and 75% following a TVM. The TVM operation is the study population that is compared to the laparoscopic CSP performed in two different technique (see methods).

The statistical power is based on a non-inferiority assumption with a binary outcome. On the basis of previous studies we estimated that 96 patients are needed in each group for 80% power to detect a 20% difference in the primary outcome measure, with a two-tailed error of 1%.

A drop-out ratio of 10% is assumed and 106 women are needed in each group (transvaginal mesh, laparoscopic colposacropexy type A and laparoscopic colposarcopexy type B). Thus, a total of 318 women are planned to be randomized for the study.

Subjective outcome:

Symptom spesific: Pelvic floor Distress Inventory (PFDI-20), Pelvic floor Impact Questionnaire (PFIQ), Pelvic Organ Prolapse / Urinary Incontinence Sexual Questionnaire (PISQ-12) Overall quality of life: 15D and RAND-36 questionnaires Pain is evaluated by visual analogue scale (VAS; 0-10) scale. The questionnaires are filled preoperatively, and after 6 months, 12 months, and 5 years.

Objective outcome:

Evaluation of the leading part of the apical point, and anterior and posterior vaginal walls (cm in relation to the hymen level) preoperatively, and after 6 months, 12 months, and 5 years.

Peri- and postoperative (both short- and long-term) complications and possible re-operations are recorded and classified according to the Claviend-Dindo.

Operation time, hospital stay, length of sick leave and costs of medications for operation and possible complications are recorded.

Cost-effectiveness:

Direct and indirect costs cover length of operation time, length of hospital stay, needed pain medication at home, other needed medication, length of sick leave, costs of possible further outpatient department visits or hospital stay with possible re-operations.

QALY calculations are based on 15D and RAND-36 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and capability to understand the study protocol either in Finnish or Swedish.
* Objectively diagnosed symptomatic apical prolapse (leading apical prolapse (points C/D) ≥ -2) and a history of previous POP operation including hysterectomy.
* No need for any other concomitant operations except colporrhaphies and possible prophylactic salpingo-oophorectomy in CSP groups

Exclusion Criteria:

* A history of serious or prolonged pain after any operation or current or previous prolonged (over 6 months) pain of any reason.
* BMI over 40
* Regular use of systemic corticosteroid medication.
* Incapability to understand the study protocol.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Subjective success; defined as the absence of vaginal bulge | 5 years
  Negative response to PDFI-20, question 3, at one-year following the surgery

SECONDARY OUTCOMES:
Peri and post-operative complications | 1 year
  peri- and post-operative complications as recorded in medical charts
Post-operative pain | 1 year
  Pain is evaluated by visual analogue scale (VAS; 0-10) scale
Objective efficacy | 1 year
  simplified POP-Q
Re-operation rate | 1 year
  re-operations
Cost-effectiveness | 1 year
  Studied by comparing both direct costs and QALYs.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki Naistenklinikka, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No